CLINICAL TRIAL: NCT01574105
Title: Heparin Dose and Post Operative Bleeding in Cardiopulmonary Bypass Patients
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Mark Rosin, Senior Clinical Perfusionist, University of Saskatchewan
Other Study IDs: 12-37
Record Dates: First submitted 2012-03-06; First posted 2012-04-10 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Disease
Keywords: Heparin Dose; Heparin Resistance; Chest Tube Losses; Transfusion Events
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Heparin Resistant: Patient whose slope calculated by a heparin dose response test is 89 sec/iu/ml or less.
- Heparin Sensitive: Patient whose slope calculated by a heparin dose response test is 90 sec/iu/ml or more.

SUMMARY:
Blood is anticoagulated using a drug named heparin during open-heart surgery to allow it to safely pass through the heart-lung machine which pumps the blood throughout the body during the surgery. Each patient is given the heparin they need for their surgery. This means some patients receive more or less heparin than other patients. In this study, the investigators will be evaluating the current anticoagulation protocol for open heart surgery in use at the Royal University Hospital. The goal of this project is to compare patients who require and receive more heparin for proper anticoagulation to those patients who require and receive less heparin.

Open-heart surgery will proceed according to the standard hospital protocol. All research participants will be treated according to standard post-open heart surgery protocol in the ICU. This will include measurement of blood loss by keeping track of chest tube outputs and administration of blood transfusions.

This study focuses on Saskatoon Health Region patients having open heart surgery in terms of the protocol for anticoagulation and blood transfusions.

DETAILED DESCRIPTION:
This study examines heparin doses of patients having cardiopulmonary bypass supported surgery in terms of their sensitivity and resistance to heparin which is the standard anticoagulant used. The investigators use the Heparin Management System, an analyser that performs a heparin dose response test. In this test, a patient's whole blood is mixed with increasing amounts of heparin to determine the required dose to achieve a set level of anticoagulation. Patients who are found to resistant to heparin and needing a higher dose are thought by some to bleed more post operatively. It is my view that when the patient is given the correct amount of heparin which is then reversed by the correct amount of protamine (the reversal agent) the bleeding is not determined by heparin dose.

Hypothesis statement: Higher doses of heparin do not cause increased postoperative bleeding and transfusion events in the postoperative CPB patient.

Purposes of the Study

1. Compare heparin sensitive and resistant patients in terms of postoperative bleeding and transfusion events.
2. Determine the incidence of heparin sensitivity or resistance in patients.
3. Identify preoperative factors that lead to heparin resistance or sensitivity in patients.
4. Using the Heparin Dose Response test in determining heparin resistant and sensitive patients.
5. Examination of anticoagulation protocol for open-heart surgery.
6. Effect of preoperative antiplatelet and anticoagulant therapy on perioperative care.
7. Use routine laboratory tests and values as well as common clinically available values in the conduct of the study so that results would be clinically relevant.

This is a prospective observational study. Patients will be divided into two groups dependant upon the results of their heparin dose response test; sensitive or resistant. Two groups of thirty will be selected to achieve 90% power at the 0.025 level of significance using a one-sided two-sample t-test.

The primary investigator will collect all data and submit the means to the statistician. Based on anecdotal experience the investigators expect there will be no difference between the two groups in terms of chest tube losses and transfusion events post-operatively.

This work is quite relevant to the investigators daily practice. Every open heart patient is anticoagulated with heparin and bleeds post operatively. The investigators goal is a reproducibly safe anticoagulation level and an acceptable level of chest tube losses. This translates to getting patients out of the operating room in a timely fashion and minimizing transfusion events.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective or urgent CABG of two to six vessels.

Exclusion Criteria:

* Preoperative:
* Hemoglobin of less than 110grams/Litre
* Under 18 years of age
* Mass less than 75 kilograms
* Presence of an intra-aortic balloon pump
* Emergency surgery, requiring operative intervention within 24 hours of consultation to the cardiac surgery team
* Need for cardiac surgical intervention in addition to planned CABG (with the exception of patent foramen ovale closure)
* Ejection fraction of less than 50%, as determined by echocardiogram or angiography
* Pulmonary hypertension with pulmonary artery pressures greater than 60mmHg
* Presence of infectious endocarditis
* Hepatic failure with impaired liver function, including INR greater than 1.5 Known diagnosed bleeding disorder
* History of heparin induced thrombocytopenia and thrombosis
* Renal failure with pre-operative creatinine greater than 200ml/min or oliguria with urine output less than 10millilitres/hour
* Allergy to tranexamic acid
* Pregnancy

Intraoperative:

* Discovery of infectious endocarditis
* Need for cardiac surgical intervention in addition to planned coronary CABG

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: On the date of surgery, the patient would be brought to the operating room. The first blood sample would be drawn prior to heparinization. This would include analysis for Activated Clotting Time, Heparin Concentration/Heparin Dose Response, antithrombin and Thrombelastograph. During this first sampling interval, the patient's Heparin Sensitivity or Resistance is determined by Heparin Dose Response (slope). The following values would determine which one of the two study groups the patient would be assigned:
  * Sensitive to heparin: at or above 90 seconds/unit/millilitre
  * Resistant to heparin: below 89 seconds/unit/millilitre
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Rosin, MPS, Principal Investigator — Saskatoon Health Region
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Began May 1, 2012 Completed January 15, 2013 Patients identified in preadmission clinic or ward.
Pre-assignment Details: Exclusion criteria included: renal failure, liver dysfunction, baseline INR >1.5, clotting factor deficiencies, intra-aortic balloon pump therapy, emergency surgery, pregnancy, ejection fraction less than 50%, age less than 18 years, pulmonary hypertension infectious endocarditis, and history of heparin induced thrombocytopenia.
Groups:
- Heparin Resistant: Patients whose heparin dose response slope was 89 sec/iu/ml or lower prior to surgery.
- Heparin Sensitive: Patients whose heparin dose response slope was 90 sec/iu/ml or higher prior to surgery.
Period: Overall Study
Arm/Group | Heparin Resistant | Heparin Sensitive
Started | 29 | 37
Completed | 29 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heparin Resistant | Heparin Sensitive | Total
Number analyzed (Participants) | 29 | 37 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 16 | 27
  >=65 years | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.8) | 67.8 (9.4) | 67.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 26 | 32 | 58
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 37 | 66

OUTCOME MEASURES:

1. Primary Outcome: Chest Tube Losses
Description: Chest tube losses will be measured in millilitres upon arrival in the Intensive Care unit (ICU) after six hours in the ICU and total chest tube losses during the ICU stay. Chest tube losses are the amount of blood collected in a graduated chest tube collection reservoir from chest tubes placed in the patient's chest wound at the end of surgery.
Time Frame: Chest tube losses are recorded from departure from operating room to chest tube removal in the ICU (normally less than 24 hrs)
Measure: Mean (Standard Deviation); unit: millilters
Arm/Group | Heparin Resistant | Heparin Sensitive
Number analyzed (Participants) | 29 | 37
millilters | 726 (371) | 781 (320)
Statistical Analysis 1: Comparison: Heparin Resistant vs Heparin Sensitive; For the analysis of the patient characteristics Wilcoxon, Chi-square and Fischer's exact tests were used. An upper bound of a two-sided 95% confidence interval (CI) of the mean difference between resistant and sensitive groups for all values of chest tube losses was computed by analysis of covariance (ANCOVA), and compared with pre-specified noninferiority limits. Covariates in the ANCOVA model included patient characteristics differing between two groups with a p-value <0.1; Test type: Non-Inferiority or Equivalence — Sample sizes of 26 in heparin resistant group and 26 in heparin sensitive group achieve 90% power at the 0.025 level of significance to detect a non-inferiority using a one-sided two-sample t-test, assuming a noninferiority margin is 200 milliliters in the postoperative chest tube loss; p < 0.1, ANCOVA

2. Secondary Outcome: Transfusion Events
Description: Transfusion events to recorded will be the number of patients receiving units of red blood cells, units of platelets, units of plasma and units of cryoprecipitate.
Time Frame: Data collection begins with patient arrival in the operating room and ends with discharge from the ICU (normally less than 24hrs)
Measure: Number; unit: Participants
Arm/Group | Heparin Resistant | Heparin Sensitive
Number analyzed (Participants) | 29 | 37
Participants | 4 [0.02 to 0.58] | 16 [0.02 to 0.58]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Heparin Resistant | Heparin Sensitive
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/37
Other Adverse Events (participants affected / at risk) | 0/29 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No